CLINICAL TRIAL: NCT03157947
Title: Development and Testing of a Culturally Tailored Decision Aid for Hispanic Patients Diagnosed With Prostate Cancer
Brief Title: Culturally Tailored Decision Aid for Hispanic Patients Diagnosed With Prostate Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study Team did not respond to requests for continuing review approval.
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE1817
Record Dates: First submitted 2017-05-16; First posted 2017-05-17 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Prostate Cancer
Keywords: decision aid; focus group
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Decision Aid (Experimental): Subjects will be asked to complete baseline surveys. Once the surveys are completed, subjects will review the Decision Aid tool with a study team member. Once the subjects have gone through the tool, study team members will answer any additional questions he may have regarding the tool. The subjects will then discuss with the investigator various cancer management options, quality of life implications, and any questions the subjects may have regarding cancer management options. Subjects that are ready may make a cancer management decision at this time, or choose to wait until their next scheduled visit. Subjects will be followed at subsequent urology clinic visits for up to 6 months. Subjects will complete follow-up surveys at the 3, 6, 9 and 12 month visits.
  Interventions: Behavioral: Decision Aid Tool; Behavioral: baseline survey; Behavioral: follow-up surveys

INTERVENTIONS:
Behavioral: Decision Aid Tool — Subjects will be given an I-pad with the decision aid program on it. A member of the study team will enter some preliminary information, then the subject will be able to review the tool with his doctor.
Behavioral: baseline survey — patients will be given baseline surveys to gather demographic information and readiness to make a decision regarding prostate cancer care
Behavioral: follow-up surveys — at 3, 6, 9, and 12 months patients will be given follow-up surveys regarding prostate cancer care

SUMMARY:
A pilot study testing the effect of an in-visit English and Spanish language decision aid for Hispanic-Latino men using best practices of cultural tailoring to be used in urology practice. Subjects will be followed for approximately 1 year during standard care in-clinic office visits. Study results and subject surveys will be analyzed to determine clinical utility of the tool.

DETAILED DESCRIPTION:
The objective of this research is to determine the effect of a culturally tailored decision aid tool on the cancer treatment decisions of Hispanic-Latino patients.

The specific aims are:

i. To develop and pilot test in an uncontrolled fashion an in-visit English and Spanish language decision aid for Hispanic-Latino men using best practices of cultural tailoring to be used in urology practice ii. To pilot and test the impact of a culturally tailored, English and Spanish language version of the Prostate Choice in-visit decision aid on decision quality, knowledge, and quality of life in low-income Hispanic/Latino patients diagnosed with localized prostate cancer iii. To assess the barriers and facilitators of decision aid use including the relative contribution of language-concordance on 1-year practice implementation parameters.

ELIGIBILITY:
Inclusion Criteria:

* Subjects utilize English or Spanish as their primary spoken or written language and identify with a Latino ethnicity and/or culture
* Men with a new histologic diagnosis of localized prostate cancer
* PSA level of 0.1 - 50 ng/dl
* Gleason score of 6 - 10
* Cancer stage: T1 - 4N x M0

Exclusion Criteria:

* Metastatic disease, including lymph nodes or distant metastasis
* PSA > 50 ng/dl
* Individuals with a medical condition that necessitates a specific prostate cancer treatment plan
* Individuals that are unwilling or unable to attend study visits or are planning to move out of a study site coverage area during the subject's anticipated participation in the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Decision Quality of cancer care in low-income Hispanic/Latino patients diagnosed with localized prostate cancer | Up to 12 months
  Decisional quality will be measured by the O'Connor Decisional Conflict Scale
Knowledge of prostate cancer care in low-income Hispanic/Latino patients diagnosed with localized prostate cancer | Up to 12 months
  Prostate cancer knowledge will be measured by the Knowledge Measurement Tool
Patient satisfaction in low-income Hispanic/Latino patients diagnosed with localized prostate cancer | Up to 12 months
  Patient satisfaction will be measured by the CAPSURE (Cancer of the Prostate Strategic Urologic Research Endeavor) patient satisfaction measurement tool

SECONDARY OUTCOMES:
Quality of Life in low-income Hispanic/Latino patients diagnosed with localized prostate cancer | Up to 12 months
  Health-related quality of life will be measured by the EPIC (Expanded Prostate Cancer Index Composite) assessment tool

CONTACTS AND LOCATIONS:
Overall Officials: Simon P Kim, MD, MPH, Principal Investigator — University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center